CLINICAL TRIAL: NCT05803889
Title: Characterization and Kinetic of Chemotherapy-induced Cardiovascular Toxicity in Breast Cancer - PROTECT-COEUR
Brief Title: Characterization and Kinetic of Chemotherapy-induced Cardiovascular Toxicity in Breast Cancer
Acronym: PROTECT-COEUR
Status: Terminated | Type: Observational
Why Stopped: The PROTECT-COEUR study had to be stopped primarily due to logistical constraints.
Sponsor: Institut de cancérologie Strasbourg Europe (Other)
Collaborators: UR 3072 (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2022-017
Record Dates: First submitted 2023-03-22; First posted 2023-04-07 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- EC + Tax group: For the EC + Taxol arm, patients will have five visits during (neo)adjuvant chemotherapy: before the start of chemotherapy (evaluation 1), before the second EC administration (evaluation 2), before the third EC administration (evaluation 3), at the end of EC sessions and before the start of Tax (evaluation 4), and at the end of Tax administration (end of chemotherapy) (evaluation 5).
  Interventions: Other: Cardiac evaluation
- Trastuzumab group: Patients in the Trastuzumab arm will be assessed only once at the end of treatment (on the same evaluation as the CE + Tax arm) to allow comparison with the fifth evaluation in the CE + Tax arm.
  Interventions: Other: Cardiac evaluation

INTERVENTIONS:
Other: Cardiac evaluation — In order to obtain information on the body composition of the patients, a body composition measurement will be performed. A resting cardiac echocardiography will be performed to record myocardial deformations in a non-vulnerable way. A non-invasive evaluation of arterial function will be performed by ultrasound on the femoral artery during a standardized passive movement of the leg. An assessment of myocardial deformations will also be performed under submaximal exercise conditions (at a target heart rate of 120 beats per minute, low to moderate exercise intensity). All of these measurements will be performed during evaluation 1 and reproduced in the same way during the 4 other sessions planned during (evaluation 2, 3 and 4) and after the treatment (evaluation 5).
  Groups: EC + Tax group
Other: Cardiac evaluation — The same measurements as the EC + Tax group will be performed but only once, at the end of the treatment.
  Groups: Trastuzumab group

SUMMARY:
The combination of epirubicin-cyclophosphamide (EC) and paclitaxel (Tax) is one of the main chemotherapy treatments used in breast cancer patients. These treatments, which can be combined with anti-HER2 therapy using trastuzumab, are frequently associated with side effects including cardiac toxicity. However, this cardiac toxicity has only been demonstrated several months after treatment and using global indices such as ejection fraction.

The assessment of myocardial dysfunction using regional deformations and the kinetic of this dysfunction during chemotherapy treatment has never been performed. In order to counteract these myocardial dysfunctions, it is essential to better describe the kinetic of the cardiac toxicity by initiating measurements since the beginning of the treatment, in order to be able to propose adapted countermeasures (e.g. exercise training) in parallel with the chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

Epirubicin-cyclophosphamide + paclitaxel group:

* Female ≥ 18 years
* Stage I to III breast cancer
* Patient being planned for (neo)adjuvant therapy combining EC and Taxol on a weekly basis
* Enrolled in a social security plan
* Able to speak, read and understand French

Trastuzumab group:

* Female ≥ 18 years of age
* Stage I to III breast cancer
* Patient treated with trastuzumab
* Enrolled in a social security plan
* Able to speak, read and understand French

Exclusion Criteria:

For both groups: Epirubicin-cyclophosphamid + paclitaxel group and trastuzumab group

* Implantation of a pacemaker
* Contraindications to exercise
* Protected adult
* Psychiatric, musculoskeletal or neurological problems
* Pregnant or breastfeeding woman
* Uncontrolled high blood pressure
* Body Mass Index > 35 kg/m²

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Population composed of a group of breast cancer patients undergoing chemotherapy with EC and Tax, and a group of breath cancer patients undergoing Trastuzumab treatment.
Sampling Method: Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2023-09-21 (Actual); Primary Completion 2024-02-15 (Actual); Study Completion 2024-02-15 (Actual)

PRIMARY OUTCOMES:
Studying the impact of chemotherapy combining EC and Tax on myocardial deformations (at rest and at submaximal effort) in order to identify the kinetic of systolic and diastolic dysfunctions. | During the treatment period, approximately 16 to 21 weeks
  Characterizing the alteration of global longitudinal strain (GLS) by resting echocardiography at rest before, during, and after chemotherapy in a group of breast cancer patients receiving EC and Tax.

SECONDARY OUTCOMES:
Studying the kinetic of the development of vascular dysfunction in order to understand a potential vascular dysfunction that could occur during treatment with chemotherapy combining EC and Tax. | During the treatment period, approximately 16 to 21 weeks
  Analyze changes in myocardial deformations during submaximal exercise, vascular function assessed non-invasively by femoral artery ultrasound, and changes in the presence of markers of myocardial injury in the blood compartment.
To compare myocardial deformations (at rest and under submaximal stress) between patients treated with EC + Tax to patients treated with trastuzumab. | During the treatment period, approximately 16 to 21 weeks
  Comparison of myocardial deformations changes induced by two types of treatment: EC + Tax and Trastuzumab. For this endpoint, we will compare the end of chemotherapy treatment to the end of trastuzumab treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Institut de cancérologie Strasbourg Europe, Strasbourg, France, France